CLINICAL TRIAL: NCT04018586
Title: AVACEN Treatment Method on Fasting and Postprandial Blood Glucose
Brief Title: AVACEN Hand Heating on Fasting Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeff Moore (Other)
Responsible Party: Sponsor-Investigator, Jeff Moore, Investigator, San Diego State University
Organization: San Diego State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AVACENFBG
Record Dates: First submitted 2019-07-06; First posted 2019-07-12 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Hyperglycemia; Hypertension
MeSH Terms: conditions — Hyperglycemia; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Heat and Vacuum (Experimental): AVACEN 100 device applies heat and vacuum to hand
  Interventions: Device: AVACEN 100
- Heat Only (Active Comparator): AVACEN 100 device with heat only
  Interventions: Device: AVACEN 100 Heat Only
- Sham (Sham Comparator): AVACEN 100 device with neither heat nor vacuum
  Interventions: Device: AVACEN Sham

INTERVENTIONS:
Device: AVACEN 100 — AVACEN 100 pulls a -30mmHg vacuum around hand from wrist down and applies heat (108 farenheit) to the palm and will be applied for 30 minutes
  Arms: Heat and Vacuum
Device: AVACEN 100 Heat Only — AVACEN 100 applies heat (108 Fahrenheit) to the palm and will be applied for 30 minutes
  Arms: Heat Only
Device: AVACEN Sham — AVACEN 100 neither heats nor pulls a vacuum to hand
  Arms: Sham

SUMMARY:
A double-blind crossover randomized controlled trial to investigate the effects of the AVACEN device on fasting blood glucose. The AVACEN device creates negative pressure around the hand while heating the palm. Two sham devices, one providing heat but no vacuum and one providing neither heat nor vacuum were also used. Each subject was tested while using each of these three devices on separate visits. Subjects arrived in the morning following an overnight fast. Fasting blood glucose, blood pressure, tympanic temperature, and subjective thermal ratings were measured before and throughout the 30 minutes that the device was used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diabetes diagnosis, diabetes medication, blood pressure medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | 30 minutes
  Change in fasting blood glucose after 30 minutes of use of AVACEN device

SECONDARY OUTCOMES:
Blood Pressure | 30 minutes
  Change in blood pressure after 30 minutes of use of AVACEN device
Tympanic Temperature | 30 minutes
  Change in tympanic temperature after 30 minutes of use of AVACEN device
ASHRAE 7 point thermal sensation scale | 30 minutes
  Change in subjective temperature after 30 minutes of use of AVACEN device

CONTACTS AND LOCATIONS:
Overall Officials: Jeff M Moore, B.S./B.S., Principal Investigator — Graduate Student
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No